CLINICAL TRIAL: NCT05790044
Title: Clonidine for Intra-oral Infra-orbital Nerve Block During Pediatric Cleft Lip Revision Surgeries: Randomized Controlled Double-blind Study
Brief Title: Clonidine for Infra-orbital Nerve Block During Pediatric Cleft Lip Revision Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, RAGAA AHMED HERDAN, professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 25353465363643
Record Dates: First submitted 2023-01-31; First posted 2023-03-29 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Placebo (Active Comparator): Children will receive intra-oral infra-orbital nerve block using bupivacaine 0.2% after induction of general anesthesia and before starting surgical procedure. Total volume of 1 ml each side.
  Interventions: Drug: Bupivacaine
- Group Clonidine (Active Comparator): Children will receive intra-oral infra-orbital nerve block using bupivacaine 0.2% and clonidine 1 ug/kg after induction of general anesthesia and before starting surgical procedure. Total volume of 1 ml each side.
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Bupivacaine — intra-oral infra-orbital nerve block with bupivacaine alone
  Arms: Group Placebo
Drug: Clonidine — intra-oral infra-orbital nerve block with bupivacaine and clonidine
  Arms: Group Clonidine

SUMMARY:
Pain in children is usually an undertreated entity. Undertreating perioperative pain could lead to various metabolic, physiologic, and neurophysiological responses. The usual means of management i.e., opioids may increase the incidence of respiratory depression in this age group. Adequate postoperative analgesia in children is a vital part of perioperative care. Good pain relief minimizes oxygen requirement, reduces cardio-respiratory demands, and promotes early ambulation and recovery. Regional block given preoperatively in combination with general anesthesia provides good preemptive analgesia. It is associated with hemodynamic stability, rapid and complete recovery, and reduced analgesic requirement in postoperative period.

Type of the study: A prospective randomized controlled double-blind study.

DETAILED DESCRIPTION:
A sample of 86 undergoing cleft lip revision under general anesthesia will be needed. The sample will be randomly divided into two equal groups: Group-I (n=43) will receive total volume of 1 ml each side.of bupivacaine (0.2%) and Group II (n=43) will receive total volume of 1 ml each side.of bupivacaine (0.2%) and 1 µ/kg of clonidine.

2.4.4 -Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …): Preoperative assessment: The day prior to surgery, all patients will undergo pre-anesthetic check-up including detailed history, physical, systemic examination, and weight of the patient. All patients will be investigated for exclusion of any of the above-mentioned contraindications. Laboratory work needed will include Complete Blood Count (CBC); Prothrombin Time and Concentration (PT& PC). All children will be kept nil per mouth 6-8 h for solids and 2 h for clear liquids. No pre-medications will be given for the purpose of the study. Preparation of the patient: Written consent from parents and emergency resuscitation equipment including airway devices, pediatric advanced life support drugs will be available. Intervention: Patients will be randomly allocated into two groups of 43 patients each: Group C: Children will receive intra-oral infra-orbital nerve block using bupivacaine 0.2% after induction of general anesthesia and before starting surgical procedure. Total volume of 1 ml each side. Group B: Children will receive intra-oral infra-orbital nerve block using bupivacaine 0.2% and clonidine 1 ug/kg after induction of general anesthesia and before starting surgical procedure. Total volume of 1 ml each side.

All patients in this study will be anesthetized by the same team of anesthesiologists and operated upon by the same surgical team who will be unaware of the study medications. General anesthesia (GA) will be standardized for all patients in both groups using 100% O2 with fresh gas flow of 6 L/min and sevoflurane with increments of 1 MAC at each breath up to 8 MAC with appropriate size face mask. Parents will be allowed to be present and collaborated during face mask induction and then leave the theater when their children close their eyes. Intraoperative monitoring will include ECG, pulse oximetry, non-invasive blood pressure, capnography, and temperature. After intravenous access securing, infusion of normal saline 0.9% solution 4 ml/ kg/h starts followed by standard fluid maintenance therapy according to the patient's weight. Endotracheal intubation (RAE-ETT) with appropriate size to the patient's age will be performed after administration of 2 mg/kg propofol. After orotracheal intubation, assisted mechanical ventilation using Ayre's T- piece will be used to maintain end-tidal carbon dioxide at 35±5 mmHg. GA will be maintained with 2-3 MAC sevoflurane. Intravenous dexamethasone 0.25 mg/kg (up to a maximum of 8 mg) will be administered as prophylactic antiemetic.

For intraoral approach of infraorbital nerve block, the patient will be placed in the supine position so that the maxillary occlusal plane forms a 45-degree angle with the floor. A cotton-tipped applicator will be used to apply a topical anesthetic to the oral mucosa of the gum line above the maxillary canine. The infraorbital foramen can be approximated by having a patient look straight ahead and imagining a line down from the pupil to the inferior border of the infraorbital ridge, bicuspid teeth, and mental foramen. The inferior orbital rim will be found with the index and middle fingers of the non-injecting hand. Once it is located, the palpating finger will remain in place to prevent losing landmarks and stop the needle from entering the orbit. The cheek will be retracted with the thumb of the non-injecting hand and then the needle will be into the mucosa above the upper second bicuspid approximately 0.5 cm from the buccal surface. The needle should be directed superiority and remain parallel to the second bicuspid until it is palpated near the foramen. Before injecting the anesthetic, it is important to aspirate to ensure the needle is not within a vessel. The anesthetic will be injected into the space. It is important to avoid injecting the anesthetic into the foramen by keeping firm pressure on the inferior orbital rim with the palpating finger. Immediate complications related to regional anesthesia will be recorded: > Systemic toxicity related to local anesthetics (seizures, heart rhythm, or conduction disorder) > Bleeding at puncture site > Pupil alteration and ocular lesion Mean arterial blood pressure (MAP), heart rate (HR), arterial oxygen saturation (SpO2), and temperature will be recorded before induction of anesthesia. After endotracheal intubation, MAP, HR, SpO2, end-tidal CO2, and temperature will be measured 5 minutes and every 15 minutes until full recovery from the general anesthesia then every 15 min in the PACU for 30 minutes.

Skin incision will be made 20 minutes after infra-orbital block. An increase in HR and MAP above 20% of baseline values with skin incision will be considered as a sign of inadequate analgesia. In this case, fentanyl 1 µg/kg will be given intravenously, and the case will be excluded from the study.

Before the end of surgery, IV paracetamol 15 mg/kg will be administered. After completion of the surgical procedure, sevoflurane administration will be discontinued, and the fresh gas flow will be increased to 8 L/min with 100% oxygen. The patient will be extubated after ensuring adequate orogastric suction and patients will be transferred directly to the post anesthesia care unit (PACU) where parents are allowed to stay with their children in a quiet and warm environment without any stimulus.

The quality of analgesia will be assessed in the PACU immediately postoperatively and then at 4, 8, 12, 16, 20 and 24 hours using FLACC pain scale. The scale has five criteria that are each assigned a score of 0, 1, or 2. The scale is scored in a range of 0-10, with 0 representing no pain while 10 is the worst pain. The results of FLACC scale were interpreted as follows: 0 = Relaxed and Comfortable; 1-3 = Mild discomfort; 4-6 = Moderate pain; 7-10 = Severe pain or discomfort or both. For postoperative pain control paracetamol intravenous infusion 15 mg/kg will be given if the recorded FLACC pain score is 4 or more. Pain scores will be recorded every 10 minutes after administration of rescue analgesia to evaluate pain relief or need for further rescue analgesia. The number of children who will need postoperative rescue analgesics and the duration of analgesia that will be taken at the time when an analgesic is required will be recorded.

Postoperative vomiting episodes will be recorded and treated with intravenous ondansetron 0.1 mg/kg. Postoperative sedation will be assessed using sedation score (1. Awake and alert. 2. Sleeping but easily arouses to voice or light touch. 3. Arouses to loud voice or shaking. 4. Arouses with painful stimuli only. 5. Unarousable). Delayed complications of the blocks will be also investigated and recorded as hematoma, restricted mouth opening, vision, sensory or motor deficit, eating disorder, and local infection.

Parents will be asked to evaluate their satisfaction regarding pain control at the end of 24 h postoperatively through 5point Likert scale (1 = very satisfied, 2 = satisfied, 3 = neither satisfied nor dissatisfied, 4 = dissatisfied, 5 = very dissatisfied). Patients will be discharged from the hospital when they are pain free and there is no other medical reason to admit them to a surgical ward.

ELIGIBILITY:
Inclusion Criteria:

* Age: 1-7 years old.
* Gender: both.
* ASA physical status I-II
* Children scheduled to undergo cleft lip revision surgeries.

Exclusion Criteria:

* History of developmental delay or mental retardation, which will make observational pain intensity assessment difficult.
* Parents refusal.
* Hypersensitivity to any local anesthetics.
* Bleeding diathesis.
* Children with co-morbid conditions like congenital heart disease, respiratory pathology and central nervous system disorders.
* Skin lesions or wounds at the puncture site of the proposed block.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain score | 24 hours
  FLACC pain score as 1-3 = Mild discomfort; 4-6 = Moderate pain; 7-10 = Severe pain

SECONDARY OUTCOMES:
Heart Rate | 2 hours
  Intraoperative heart rate monitoring
Sedation Score | 6 hours
  1. Awake and alert. 2. Sleeping but easily arouses to voice or light touch. 3. Arouses to loud voice or shaking. 4. Arouses with painful stimuli only. 5. Unarousable
rescue analgesia | 24 hours
  Total rescue doses of paracetamol IV over 24 hours postoperatively used in each group.
5-point Likert scale Satisfaction Score | 24 hours
  1 = very satisfied, 2 = satisfied, 3 = neither satisfied nor dissatisfied, 4 = dissatisfied, 5 = very dissatisfied

CONTACTS AND LOCATIONS:
Overall Officials: Ragaa Herdan, professor, Principal Investigator — faculty of medicine assiut university egypt

IPD SHARING:
Plan to Share IPD: No